CLINICAL TRIAL: NCT03302949
Title: Nutritional Supplement Trial in Patients With Tuberculosis to Improve Anthropometry and Treatment Outcome
Brief Title: Treating Tuberculosis Wasting With a High-protein Supplement
Acronym: NUTRIATO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment stopped before reaching sample size due to time constraints. Follow up visits and intervention was given per protocol to all included participants.
Sponsor: University of Aarhus (Other)
Collaborators: Bandim Health Project (Other); Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1004
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Undernutrition; Malnutrition
Keywords: Nutritional Supplement; Health-related Quality of Life; Dietary Intake
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control arm will not receive the intervention, but will receive standard 6-month anti-tuberculosis regimen and nutritional supplements provided by various NGO's (on irregular basis).
- Intervention (Experimental): Intervention arm will receive standard 6-month anti-tuberculosis regimen, nutritional supplements provided by various NGO's (on irregular basis), and receive the study intervention of daily supplement of 62.5g Lacprodan® DI-8090
  Interventions: Dietary Supplement: Lacprodan® DI-8090

INTERVENTIONS:
Dietary Supplement: Lacprodan® DI-8090 — Whey protein concentrate. 100g powder contains 392 kcal (1646 kJ), hereof 80% protein.
  Arms: Intervention

SUMMARY:
Undernutrition at the time of diagnosis of active tuberculosis is a risk factor for increased mortality, and lack of weight gain during anti-tuberculous treatment has been linked to an increased relapse risk. The purpose of this study is to test the effect of Lacprodan® DI-8090 whey protein concentrate on anthropometric measures, treatment outcome and health-related quality of life, against standard practice during anti-tuberculous treatment on patients with a BMI <20 living in Guinea-Bissau.

DETAILED DESCRIPTION:
It is hypothesized that patients with tuberculosis receiving whey protein concentrate as nutritional supplement will experience a greater gain in adverse anthropometric measures, and experience a decreased risk of relapse and death, compared with patients with tuberculosis, who do not receive nutritional supplement. 260 patients will be recruited from and included/randomized at 4 trial sites in Bissau, Guinea-Bissau (Bandim Health Center, Belem Health Center, Cuntum Health Center and Hospital Raoul Follereau). Patients randomized to the intervention arm will receive one package of whey protein concentrate (approx. 62.5g) per day for the duration of the 6-month long anti-tuberculous treatment. Patients will be followed bimonthly during the treatment period, with clinical examinations, blood sample analyses, and nutritional status and dietary intake assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with TB
* Aged 18 years and above
* BMI<20

Exclusion Criteria:

* Pregnancy
* Commencement of treatment ≥30 days prior to inclusion
* Decreased kidney function
* Missing informed consent
* Mentally ill/disabled patients unable to comply with the treatment/intervention regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Anthropometry | 6 months
  Proportion of patients with BMI gain >9% at end of treatment

SECONDARY OUTCOMES:
Treatment Outcome | 6 months
  Defined by WHO criteria (incl. mortality), at end of treatment
Treatment outcome | 2 years
  Defined by WHO criteria (incl. mortality), at 2-year follow up
Anthropometry | 2 years
  Proportion of patients with sustained BMI gain >9% at 2-year follow up
Diet | 6 months
  Assesment of daily energy intake (kJ) of patients with tuberculosis using sq-FFQ
Health-related quality of life | 6 months
  Score obtained from SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie B Patsche, Principal Investigator — University of Aarhus
Locations (1):
- The Bandim Health Project, Bissau, Denmark, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No